CLINICAL TRIAL: NCT04434326
Title: A Single-center, Open-label, Single-dose Phase I Study to Investigate the Absorption, Metabolism and Excretion of [14C]CM082 After a Single Oral 200mg/100µCi Dose in Healthy Chinese Male Subjects
Brief Title: The Absorption, Metabolism and Excretion of [14C]CM082 in Human
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AnewPharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM082-CA-I-109
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2021-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]CM082 (Experimental): To investigate the absorption properties, as well as to evaluate the mass balance and elucidate the pathways of biotransformation after a single oral dose (200mg, 100µCi) of [14C]CM082 to healthy Chinese male subjects
  Interventions: Drug: [14]CM082 suspension

INTERVENTIONS:
Drug: [14]CM082 suspension — Before administration, the solid powder for administration was placed at room temperature. 40 ml drinking water was added into the drug container to prepare the suspension for the subjects to take. After that, 200 ml drinking water was used to repeatedly rinse the drug container for many times, and the subjects continued to take the lotion. Take care not to spill the liquid out of the bottle when shaking

SUMMARY:
This is a single-center, open-label, single-dose phase I study to investigate the absorption, metabolism and excretion of [14C] CM082 in healthy Chinese male subjects. The study will be conducted into two steps：Firstly, 2 subjects are enrolled in to participate in the pilot study to grope for the completion date of plasma, urine and feces sampling on the 3rd day post-dose and onwards. Then, the collection time of blood and excreta samples (urine and feces) from the subsequent 4-6 subjects will be adjusted according to the pilot study

DETAILED DESCRIPTION:
Subjects who had signed informed consent and meet inclusion criteria and no exclusion criteria are admitted to Phase I Clinical Unit two days prior to dosing (D-2). On the morning of Day 1 before dosing, subjects will be transferred to nuclear medical ward. And after an overnight fast of at least 10 h, subjects will receive a single oral dose of 200 mg (100 μCi) of [14C]CM082 as an oral suspension. Then, after two days of the dosing, subjects will be transferred back to Phase I Clinical Unit ward and confined to this unit until blood or excreta sampling and safety monitoring at the designated time points or intervals are complete

ELIGIBILITY:
Inclusion Criteria:

* 1.healthy male volunteers between the ages of 18 to 50 years old; 2.Body weight >=50 kg, Body mass index (body weight(kg)/hight2(m2)) between 19 and 26 kg/m2; 3.Normal physical findings, clinical laboratory values, vital signs and 12-lead ECG, or any abnormality that is non-clinically significant; 4.Male subjects of reproductive potential with partners will be instructed to, and must be willing to practice a highly effective method of birth control for the duration of the study and continuing 1 year after discontinuing treatment with the investigational product. Highly effective methods of birth control include using condom, contraceptive sponge, contraceptive gel, contraceptive film, intrauterine device, oral or injectable contraceptive pill, hypodermic implants or others; 5. Must understand, and voluntarily sign the informed consent, comply with the requirements of the study.

Exclusion Criteria:

* 1.History of or current clinically significant cardio, pulmonary, endocrine, metabolism, renal, hepatic, gastrointestinal, dermatology, infection, hematology, neurological, mental disease or disorder; 2.Positive test for HBsAg, HBeAg, anti-HCV, anti-HIV or syphilis antibody; 3.History of syncope / needle syncope and intolerable intravenous indwelling needle; 4.History of clinically significant disease or infection within 1 month before entering the study; 5.Abnormality in blood pressure, including hypertensive BP (SBP>=140 mmHg, or DBP >=90 mmHg), or hypotensive BP(SBP<90 mmHg, or DBP <=55 mmHg), Pulse rate<55 bpm or >100 bpm; 6.Long-QT syndrome or family history of it, or QTcB interval > 450 ms; intraventricular blocks or left/right bundle branch block or QRS>120ms; frequent ventricular ectopic beats (any 10s ECG ventricular premature beat >= 1 in screening period); or abnormal resting heart rate (> 100 bpm); 7.The following abnormal clinical laboratory values

  1. HGB < LLN, and is judged as clinically significant by the investigator；
  2. Abnormal ALP, ALB,TP,Cr,ALT,AST,BIL,Urea, GLU value, and is judged as clinically significant by the investigator; 8.Received any drug within 14 days before taking the investigational drug, including any prescription drug, OTC drug, herbal drug or health care products, except for vitamins and paracetamol； 9.History of or current swallowing disorder, active gastrointestinal diseases, or other diseases that significantly affect absorption, distribution, metabolism and excretion of drugs; 10.Chronic constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease; 11.Hemorrhoids or perianal disease with regular/perianal bleeding; 12.Allergies, have allergies to two or more drugs or foods; or have known allergies to the components of the drug (Mannitol, sodium bicarbonate, sodium dodecyl citrate, sodium carboxymethylcellulose, povidone, silica, magnesium stearate); 13.Have donated 500ml or more of blood or plasma 2 months prior to the study drug administration, or more than 50ml within 2 weeks prior to administration; 14.Vaccination was administered within 6 months prior to screening or during screening; 15.History of drug or alcohol abuse; 16.Smoking (> 10 cigarette / day), drinking (> 15 g, pure alcohol / day, equivalent to 450 ml beer, 150 ml wine or 50 ml low-alcohol liquor), or abusing drugs(MOP, METmAMP, MTD, THC, AMP positive) within last 3 months; 17.Subject with mentally ill and could not understand the property, scope and possible consequences of the study; 18.subject in prison or whose freedom is restricted by administrative or legal issues; 19.Failure to comply with clinical study protocols, such as non-cooperation, follow-up visit and completion of entire study; 20.Investigator, pharmacist, CRC or research associate; 21.Participated in other clinical trials within 3 months before screening; 22.The subjects participated in the clinical trial of radioactive labeling within one year before taking the medicine; 23.Significant radiation exposure within one year prior to drug administration (more than one exposure from chest X-ray, CT scan, or barium meal examination and radiation-related occupations); 24.Investigators think that subjects are not suitable to participate in the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2021-10-22 (Actual)

PRIMARY OUTCOMES:
Radioactivity concentration of each plasma sample | Day 1-Day6
  Use liquid scintillation counter to evaluate Radioactivity concentration of each plasma（DPM/ml) sample
Radioactivity concentration of each urine samples | Day-1-Day11
  Use liquid scintillation counter to evaluate Radioactivity concentration of each urine（DPM/ml） sample
Radioactivity concentration of each feces sample | Day-1-Day11
  Use liquid scintillation counter to evaluate Radioactivity concentration of each feces（DPM/g） sample
Total recovery of radioactivity in urine and feces | Day-1-Day11
  Calculate the total radioactivity in urine and feces based on the radioactivity concentration of each sample.
Identification of metabolites in plasma, urine and fecal samples | Day-1-Day11
  LC-MS was used to identify the main metabolites in plasma, urine and feces, and finally to provide the main biotransformation pathway of CM082 in human body

SECONDARY OUTCOMES:
Plasma drug concentrations | Day-1-Day11
  To determine the plasma concentrations of CMO82 with validated LC-MS/MS method for obtaining its pharmacokinetics parameters
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | Day-14-Day11
  According to CTCAE v4.03, the number and frequency of adverse events after a single dose of test drug were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shao, Ph D, Principal Investigator — Jiangsu Province Hospital Affiliated to Nanjing Madical University of Medicine; Wei Liu, M.A, Principal Investigator — Jiangsu Province Hospital Affiliated to Nanjing Madical University of Medicine
Locations (1):
- Jiangsu Province Hospital Affiliated to Nanjing Madical University of Medicine, Nanjing, Jiangsu, China